CLINICAL TRIAL: NCT03238989
Title: Interstitial Lung Disease Registry Construction
Acronym: ILD Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sun Mi Choi, Assistant professor, Seoul National University Hospital
Other Study IDs: ILD Registry
Record Dates: First submitted 2017-07-27; First posted 2017-08-03 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Interstitial Lung Disease
Keywords: Interstitial lung disease
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: monitoring changes in clinical symptoms, pulmonary function, and chest radiography — For patients with interstitial lung disease, the investigators regularly monitor changes in clinical symptoms, pulmonary function, and chest radiography after basic questionnaire on symptoms, lifestyle, depression, and quality of life.

SUMMARY:
The purpose of this study is investigating the clinical course, treatment course, and prognosis of patients with interstitial lung disease.

DETAILED DESCRIPTION:
Interstitial lung disease refers to pulmonary disease that occurs in the interstitium of the lung.

It can be broadly classified into lung disease secondary to the cause of systemic disease or drug, and lung disease whose cause is unknown, and the latter is known as idiopathic interstitial pneumonia.

Idiopathic interstitial pneumonia is a lung disease showing various aspects of inflammatory response and fibrosis reaction, and the cause of the onset is not accurately known yet, also there is no effective treatment.

Idiopathic interstitial pneumonia, including idiopathic pulmonary fibrosis, progresses very slowly, but sometimes acute exacerbation without any obvious cause leads to death, rapidly.

Therefore, it is important to collect data prospectively for changes in clinical features, pulmonary function, imaging findings, and quality of life of these patients.

A prospective study of idiopathic interstitial pneumonia will provide important information on the clinical characteristics and admission history of patients with idiopathic interstitial pneumonia, and the idiopathic interstitial pneumonia registry system will serve as the basis for further prospective observational studies.

The aim of this study is to establish the registry of patients with interstitial lung disease and to prospectively review the clinical features and progression of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 20 years diagnosed with interstitial lung disease
* Diagnostic criteria for interstitial lung disease. If one of the following is met:

  1. clinical suspicion of idiopathic pulmonary fibrosis (IPF); Characteristic chest CT findings with honeycomb cysts and fibrosis and reasonable clinical signs
  2. suspected interstitial pneumonia, or confirmed by biopsy with no evidence of infection : IPF, Non-specific interstitial pneumonia(NSIP), Cryptogenic organizing pneumonia(COP), unclassified fibrosis
  3. interstitial lung disease suspects with underlying rheumatic disease

Exclusion Criteria:

* No specific criteria

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: outpatient, ward
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-01-05 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
St George's Respiratory Questionnaire(SGRQ) | at baseline, every 1 year through study completion for 10 years
  monitoring changes in clinical symptoms
modified Medical Research Council (mMRC) dyspnea scale | at baseline, after 1 month, after 3 month, and then every 1 year through study completion for 10 years
  monitoring changes in clinical symptoms
Borg dyspnea scale | at baseline, after 1 month, after 3 month, and then every 1 year through study completion for 10 years
  monitoring changes in clinical symptoms
Hospital anxiety and depression score(HADS) | at baseline, every 1 year through study completion for 10 years
  monitoring changes in clinical symptoms
chest X-ray | at baseline, after 1 month, after 3 month, and then every 1 year through study completion for 10 years
  monitoring changes in chest radiography
Chest CT | at baseline, every 1 year through study completion for 10 years
  monitoring changes in chest radiography
Paranasal sinus X-ray(PNS series) | at baseline
  baseline PNS X-ray
Electrocardiogram(ECG) | at baseline
  baseline ECG
Pulmonary function test with bronchodilator response test(PFT+BDR) | at baseline, after 1 month, after 3 month, and then every 1 year through study completion for 10 years
  monitoring changes in lung function
Diffusing capacity of the lungs for carbon monoxide(DLCO) | at baseline, after 1 month, after 3 month, and then every 1 year through study completion for 10 years
  monitoring changes in lung function
total lung capacity(TLC) | at baseline
  monitoring changes in lung function
Bronchoscopic alveolar lavage(BAL) | at baseline
  for diagnostic purposes if necessary
Video-assisted thoracoscopic surgery(VATS) lung biopsy | at baseline
  for diagnostic purposes if necessary
echocardiography | at baseline
  additionally tested at acute exacerbation
arterial blood gas analysis(ABGA) | at baseline
  additionally tested at acute exacerbation

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea